CLINICAL TRIAL: NCT06314841
Title: Polytrauma and Resuscitation Impact on Innate Immunity
Acronym: PRIME
Status: Terminated | Type: Observational
Why Stopped: Recruitment could not be resumed due to the COVID-19 pandemic
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Collaborators: AUVA (Other)
Responsible Party: Principal Investigator, Gerhard Fritsch, Priv.-Doz., Prim., Dr.med.univ, Ludwig Boltzmann Gesellschaft
Other Study IDs: LBG-AUVA
Record Dates: First submitted 2018-07-30; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2018-07

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral whole blood. Anticoagulants: Sodium-citrate, EDTA, Heparin. Retention of plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major trauma can lead to a dysregulated response to secondary infection. Severe injuries are accompanied by pro- and antiinflammatory changes that affect both adaptive and innate immunity. In this study we aim to assess cellular immuno-competence early during treatment in an attempt to identify signs of immuno-suppression.

DETAILED DESCRIPTION:
Polytrauma represents one of the most challenging critical conditions for caretakers worldwide and involves multiple damages of different anatomical regions. Severe traumatic injuries are among the primary causes of death among young people under the age of 45 and half of them are due to uncontrollable bleeding. In the acute injury phase of trauma, severe blood loss is often accompanied by biochemical, cellular and physiological dysfunctions leading to an inflammatory response, infections and in some cases coagulopathy. We aim to identify immuno-suppression by analyzing phagocytic capacity, leukocyte subsets, surface molecule expression and extracellular vesicles in the peripheral blood of severly injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Injury Severity Score (ISS) > 15
* Incident to admission time < 3h

Exclusion Criteria:

* Preexisting condition
* Pregnancy or breastfeeding
* Diabetes
* Coronary Heart Disease
* Intake of antiphlogistic medication
* Neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Polytraumatized patients older than 18 years, that were directly (within 3 hours) admitted to the emergency room of one the participating trauma centers and that do not match one of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Immunocompetence | 30 days after admission to ER
  Infection during observation period

SECONDARY OUTCOMES:
Changes in cellular immuno-status | 0 hours, 24 hours, 48 hours, 96 hours after admission to ER
  Flow cytometric assessment of leukocyte subsets and the expression of surface molecules involved in antigen presentation and immuno-suppression.
Release of extracellular vesicles and associated content | 0 hours, 24 hours after admission to ER
  Flow cytometric assessment of the release of extracellular vesicles from various cell types.
Platelet-leukocyte aggregates | 0 hours, 24 hours after admission to ER
  Formation of platelet-leukocyte aggregates in the peripheral blood upon admission and on the ICU.
Immunocompetence clusters | 30 days after admission to ER
  Clustering of patient immunocompetence characteristics by artificial intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Drechsler, DVM, Study Chair — Ludwig Boltzmann Institute for Experimental and Clinical Traumatology; Marcin Osuchowski, DVM, Study Chair — Ludwig Boltzmann Institute for Experimental and Clinical Traumatology; Heinz Steltzer, MD, Prof., Study Chair — Trauma Center Vienna, Meidling
Locations (3):
- Austria (3):
  - Trauma Center Vienna, Meidling, Vienna
  - Ludwig Boltzmann Institute for Experimental and Clinical Traumatology, AUVA Trauma Research Center, Vienna
  - Trauma Center Vienna, Lorenz Böhler, Vienna